CLINICAL TRIAL: NCT00495092
Title: Efficacy of Caffeine, With and Without Biperiden, in the Detoxification of Cocaine Dependent Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Miguel Casas Brugué, Servei de Psiquiatria. Hospital Universitari Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAF-DTX-1; INT/71525/2003
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Cocaine Related Disorders
Keywords: cocaine dependence; cocaine use; cocaine craving
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Caffeine; Biperiden

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): This study arm will receive caffeine+placebo
  Interventions: Drug: Caffeine
- 2 (Experimental): this study arm will receive Caffeine+Biperiden
  Interventions: Drug: Caffeine; Drug: Biperiden
- 3 (Placebo Comparator): this study arm will receive placebo+placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — Caffeine from 300 mg/d to 1200 mg/d or 15 mg/kg/d
  Arms: 1; 2
Drug: Biperiden — Biperiden 2-4 mg/d p.o.
  Arms: 2
Drug: Placebo — Placebo + Placebo
  Arms: 3

SUMMARY:
The aim of this study is to assess the efficacy of caffeine compared to placebo in detoxifying cocaine dependent patients. Caffeine potentiation with biperiden will be also studied.

108 with cocaine dependence will be randomized to receive caffeine (300 - 1200 mg t.i.d.) plus biperidene (8 mg b.i.d.) or caffeine (300 - 1200 mg t.i.d.) with placebo or placebo during 6 months.

Primary efficacy outcomes will be 1) patient comfort assessed with abstinence symptomatology, craving for cocaine and mental status during detoxifying period, 2) study retention and 3) cocaine use.

Brain dopamine system will be assessed thru IBZM-SPECT and the apomorphine test.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of intranasal cocaine dependence, according to DSM-IV-TR criteria
* age between 18 and 60 years
* current cocaine use, confirmed by a positive urine drug screen for cocaine the week prior to admission.
* demonstrated capacity to grant informed consent and sign the pertinent informed consent form.
* place of residence compatible with attendance at the centre.
* for women, willingness to use effective contraceptive measures during the study.

Exclusion Criteria:

* diagnosis of a severe medical disorder that could interfere with the study
* presence of an organic pathology for which methylxanthines or biperidene, iodine or apomorphine administration is contraindicated
* serum liver transaminase levels 3 times higher than normal values
* pregnancy and breast-feeding
* neuroleptic medication treatment in the past 6 weeks
* current treatment, or anticipation that the patient may need to initiate treatment during the study with drugs that may interact with study medication.
* current diagnosis of a major mental disorder.
* awareness of a situation that could prevent the patient's participation in the study (e.g. serving a sentence)
* current participation in another research project.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
1) comfort with cocaine detox defined as cocaine abstinence symptoms, cocaine craving, depressive symptoms and anxiety symptoms 2) study retention and 3) cocaine use. | 12-14 days for primary otcome num 1 and 23 weeks for num 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Casas, Prof., Principal Investigator — Hospital Universitari Vall d'Hebron Barcelona, Catalonia, Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain